CLINICAL TRIAL: NCT06574022
Title: Post-mastectomy Recovery: A Randomized Clinical Trial Comparing Preoperative PECS-II Blocks With Intraoperative Pectoral Blocks
Brief Title: Post-mastectomy Recovery: Comparing Preoperative PECS-II Blocks With Intraoperative Pectoral Blocks
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Alicia Heelan, Principal Investigator, University of Cincinnati
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: UCCC-BRE-23-01
Record Dates: First submitted 2024-08-09; First posted 2024-08-27 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Mastectomy; Lymphedema; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Bupivacaine; Operative Blood Salvage; Phenoxybenzamine

STUDY DESIGN:
Intervention Model Description: Study Design Summary:
  Stage I: A randomized trial to assess the effectiveness of AT combined with IOB.
  Stage II: Based on Stage I results, evaluate two BTs. Enroll 40 patients per group (n1 = 40, n2 = 40) to achieve 80% power at α = 0.05, with one interim analysis after 50% enrollment.
  If interim results (n1 = 20, n2 = 20) show a p-value < 0.025 when comparing pill counts (hypothesizing EX is superior to PB), proceed to Stage II. If not, continue enrollment to full sample size and reanalyze.
  If final p-value < 0.025, EX is considered superior. If not significant, continue with EX. If EX is inferior to PB, conduct subset analysis and revise inclusion/exclusion criteria for Stage II.
  In Stage II, test BT efficacy using the superior AT. Enroll 60 patients, randomized 2:1 favoring CPT. Include Stage I patients treated with IOB and superior AT in analysis. Final sample sizes: n1 = 40 or 60, n2 = 40, maintaining ≥80% power.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1) Intraoperative Pecs Blocks (IOB) & 30 cc of 0.5% bupivacaine (PB) (Active Comparator): Intraoperative direct visualization of the pectoralis nerves and injection using a 21-gauge needle of 30 cc of 0.5% bupivacaine after mastectomy completion and prior to reconstruction, if performed, or wound closure.
- 2) Intraoperative Pecs Blocks (IOB) & 20 cc of Exparel mixed w/10 cc of 0.5% bupivacaine (EX) (Active Comparator): Intraoperative direct visualization of the pectoralis nerves and injection using a 21-gauge needle of 20 cc of Exparel mixed with 10 cc of 0.5% bupivacaine after mastectomy completion and prior to reconstruction, if performed, or wound closure.
- 3) Intraoperative Pecs II block (IOB) & superior AT (EX or BP) (Active Comparator): Intraoperative direct visualization of the pectoralis nerves and injection using a 21-gauge needle with superior anesthetic as determined by stage I, after mastectomy completion and prior to reconstruction, if performed, or wound closure.
  Interventions: Procedure: Intraoperative Pecs II block (IOB) & superior AT (EX or BP)
- 4) Preoperative Pecs II block (POB) & superior AT (EX or BP) (Active Comparator): Preoperative Pecs II block to be administered by 1 of 6 acute pain specialized anesthesiologists in same day surgery. Patient will be lightly sedated with midazolam, at the discretion of the anesthesiologist. The pecs II block will be performed under ultrasound guidance using a 21-gauge, 80 mm length needle to administer the superior anesthetic as determined in stage I.

INTERVENTIONS:
Drug: Bupivacain — Intraoperative direct visualization of the pectoralis nerves and injection using a 21-gauge needle of 30 cc of 0.5% bupivacaine after mastectomy completion and prior to reconstruction, if performed, or wound closure.
Drug: Exparel — Intraoperative direct visualization of the pectoralis nerves and injection using a 21-gauge needle of 20 cc of Exparel mixed with 10 cc of 0.5% bupivacaine after mastectomy completion and prior to reconstruction, if performed, or wound closure.
Procedure: Intraoperative Pecs II block (IOB) & superior AT (EX or BP) — Intraoperative direct visualization of the pectoralis nerves and injection using a 21-gauge needle with superior anesthetic as determined by stage I, after mastectomy completion and prior to reconstruction, if performed, or wound closure.
  Arms: 3) Intraoperative Pecs II block (IOB) & superior AT (EX or BP)
Procedure: Preoperative Pecs II block (POB) & superior AT (EX or BP) — Preoperative Pecs II block to be administered by 1 of 6 acute pain specialized anesthesiologists in same day surgery. Patient will be lightly sedated with midazolam, at the discretion of the anesthesiologist. The pecs II block will be performed under ultrasound guidance using a 21-gauge, 80 mm length needle to administer the superior anesthetic as determined in stage I.

SUMMARY:
The purpose this research is to compare two different standards of care for pain management and two different standards of care for local numbing medicine for breast cancer patients who will have a total mastectomy.

DETAILED DESCRIPTION:
The purpose this research is to compare two different standards of care for pain management and two different standards of care for local numbing medicine for breast cancer patients who will have a total mastectomy.

Standard of care intervention is preoperative PECS-II blocks versus Intraoperative Pectoral Blocks.

The medication used are standard of care and include Bupivacaine and liposomal bupivacaine. Bupivacaine is FDA approved and indicated for the local or regional anesthesia or analgesia for surgery procedures and therapeutic procedures. Liposomal bupivacaine is FDA approved and indicated for adults to produce postsurgical local analgesia and as nerve block to produce postsurgical regional analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years of age or older
* Patients undergoing mastectomy with or without axillary surgery, with or without reconstruction surgery at UCMC for breast cancer or high-risk of breast cancer. Patients with high-risk of breast cancer are those who have atypical/precancerous breast lesion(s), genetic mutation with increased risk of cancer (e.g., BRCA1, BRCA2 etc..) and/or a strong family history of breast cancer in the opinion of the investigator.

Exclusion Criteria:

* Patients undergoing only a partial mastectomy or tissue-based reconstruction.
* Non-English speaking.
* Patients who are pregnant.
* Patients with an allergy to local anesthetics
* Except: patients with allergies only to topical anesthetics may be included.
* Patients with a preoperative acute or chronic pain disorder with an opioid prescription that has been prescribed within 30 days of surgery. Patients who have not filled such a prescription or who state they have not taken the medications prescribed, may be eligible on a case-by-case basis per investigator judgement.
* Patients with a history of opioid use disorder.
* Inability to provide informed consent.
* Patients who otherwise in the opinion of the Investigator are not good candidates for participation (e.g., deemed unreliable for follow-up).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain as indicated by postoperative opioid use via total inpatient and outpatient opioid use (oral morphine milliequivalents) | 14 days post-operation
  Post-operative opioid usage as measured by total inpatient and outpatient opioid use (oral morphine milliequivalents) through 14 days post-op.
Postoperative pain as indicated by postoperative opioid use discontinuation | 14 days post-operation
  Post-operative opioid usage as measured by time to opiate discontinuation through 14 days post-op.

SECONDARY OUTCOMES:
Post-operative pain scores indicated by patient report Numeric Rating Scale | 21 days Post Operation
  Post-operative pain scores as measured by the Numeric Rating Scale pain scores. Maximum, minimum, and mean pain scores on a scale of 0-10 each day of hospitalization, starting day of surgery.
Post-operative pain scores indicated by patient survey | 21 days Post Operation
  Post-operative pain scores as measured by patient survey. Patient survey completed on post-operative days 1 (while inpatient) and at their post-operative appointment (1-3 weeks post-op). The patient survey is based on the Clinically Aligned Pain Tool which is a newer tool that attempts to address some of the major limitations inherent with the much more basic numeric rating scale. A score of 1 is the minimum while a score of 10 is the maximum. The higher the score, the more pain the patient is reporting.
Patient satisfaction indicated by patient report | 21 days Post Operation
  Patient satisfaction measured at the patient's first postoperative visit (1-3 weeks post-op) using a 10-point Likert scale. The 10 Point Likert Scale will have minimum value of 1 and maximum of 10 with 1 being least satisfied (worse outcome) and 10 being most satisfied (better outcome).
Intraoperative procedure time measured as from time of incision to start of closing | Day 0: Surgery
  Total intraoperative procedure time will be measured as from time of incision to start of closing if no reconstruction is performed or to time of Panel 1 completion to be followed by the reconstruction procedure by Panel 2.
Intraoperative opioid administration measured in Milliequivalents | Day 0: Surgery
  Intraoperative opioid administration in IV Morphine Milliequivalents.
Operating room delays measured as anesthesia start time that is greater than 1 hour after the scheduled start time | Day 0: Surgery
  Number of operating room delays will be measured as anesthesia start time that is greater than 1 hour after the scheduled start time.
Postoperative length of stay as measured by the number of nights spent in the hospital after surgery. | Day 0-7
  Postoperative length of stay as measured by the number of nights spent in the hospital after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No